CLINICAL TRIAL: NCT03930303
Title: Impact of Media-based Patient Education on Anxiety Scores in Patients Undergoing Dilatation and Curettage at Office Setting
Brief Title: Anxiety Scores With Media Based Patient Education Before Dilatation and Curettage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulseren Yilmaz, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Gulseren1
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Abnormal Uterine Bleeding; Anxiety
Keywords: dilatation and curettage; multimedia based education; anxiety
MeSH Terms: conditions — Metrorrhagia; Anxiety Disorders; Dilatation, Pathologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimedia Arm (Active Comparator)
  Interventions: Behavioral: Multimedia- based patient education
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Multimedia- based patient education — Patients will receive a 5 minutes video education before D&C
  Arms: Multimedia Arm

SUMMARY:
Subjects with abnormal uterine bleeding and scheduled for dilatation and curettage (D&C) will be randomized to a multimedia-based education (MME group) or verbal information (Control group ) before (D&C). State-Trait Anxiety Inventory will be asked by the nursing staff before and after multimedia-based education or verbal information to all patients. Then the patients will undergo (D&C) at an office setting. The impact of MME on patient anxiety will be evaluated by statistical analysis.

DETAILED DESCRIPTION:
Subjects with abnormal uterine bleeding and scheduled for dilatation and curettage (D&C) with diagnostic or treatment purpose will be randomized to two intervention arms. Multimedia-education Group (MME group) and verbal information group (Control Group). Both groups will receive State-Trait Anxiety Inventory before and after education and then will undergo D&C at an office setting. State-Trait Anxiety Inventory will be asked by the nursing staff. Multimedia-based education will be carried out using a 5 minutes video explaining the details of D&C. D&C will be carried out at office setting by an experienced gynecologist under sedation and analgesia.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of abnormal uterine bleeding Scheduled for dilatation and curettage Must understand the characteristics of the study

Exclusion Criteria:

Psychological disease Contraindication for hysteroscopy Visual deficit, Auditory deficit

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change in State-Trait Anxiety Inventory score from baseline to watching video or verbal information | 30 minutes before and 10 minutes after multimedia education/verbal information
  Total score for both State anxiety inventory and Trait anxiety score (Range: 20 to 80 points, higher values represent a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Kiyak, MD, Study Chair — Kanuni Sultan Suleyman Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided